CLINICAL TRIAL: NCT06490133
Title: Nutritional Intervention to Evaluate the Effectiveness of the Consumption of Dehydrated Olive Pulp in Reducing Total Cholesterol Levels in Subjects with Overweight-obesity and High Total Cholesterol Levels
Brief Title: Evaluation of Consuming Olive Extract on Total Cholesterol Levels
Acronym: OLICOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OLICOL
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-09

CONDITIONS: Metabolic Syndrome | Serum or Plasma | Chemistry - Non-Challenge; Overweight
Keywords: polyhpenols from olives; metabolic syndrome; cholesterol; lifestyle
MeSH Terms: conditions — Metabolic Syndrome; Overweight

STUDY DESIGN:
Intervention Model Description: Parallel groups double blind, 12-week nutritional intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Capsules containing placebo.
  Interventions: Dietary Supplement: Placebo
- Polyhpenol extract (Experimental): Capsules containing the experimental polyhpenol to be assayed
  Interventions: Dietary Supplement: Polyhpenol extract

INTERVENTIONS:
Dietary Supplement: Polyhpenol extract — Three capsules in fasting conditions 15 minutes prior breakfast
  Arms: Polyhpenol extract
Dietary Supplement: Placebo — Three capsules in fasting conditions 15 minutes before breakfast
  Arms: Placebo

SUMMARY:
The main objective of this nutritional intervention is to assess the efficacy of polyphenol-rich capsules on reducing metabolic syndrome traits, mainly cholesterol levels. For this purpose, a double blind, placebo controlled study of 12 weeks will be carried out.

The target population is women and men with overweight or obesity. Researchers will compare the experimental capsules with placebo capsules, but will be blinded during the intervention and results analyses. Only after analysing the parameters, the groups will be revealed.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 35 Kg/m2
* Total Cholesterol levels in peripheral blood above or equal to 200 mg/dL or LDL-cholesterol levels above or equal to 160 mg/dL.
* Weight stability during the three months prior the start of the study (±5% of variation).
* To be able to attend the visits and accomplish with all the indications of the research staff.
* To have signed the written informed consent.

Exclusion Criteria:

* Any alteration of the Gastrointestinal system, functional or structural (gastric ulcer, chronic inflammatory diseases, hernia, etc.)
* Subjects having undergone any surgical operation in th egastrointestinal tract with permanent consequences (i.e. gastroduodenectomy).
* Subjects following any pharmacological treatment affecting gastric homeostasis.
* Suffer from any metabolic disease or cancer process.
* Being allergic to any of the compounds contained in the study capsules.
* Excessive alcohol ingestion (14 units/day for women, or 20 units/day for men).
* Women lactating or during pregnancy.
* Following any cholesterol-lowering treatment.
* People with any mental impairment or whose compliance with the study protocol is at risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-09-08 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Total cholesterol | Baseline
  Serum concentration of Total Cholesterol
Total cholesterol | 12 weeks
  Serum concentration of Total Cholesterol
HDL cholesterol | Baseline
  Serum concentration of HDL cholesterol
HDL cholesterol | 12 weeks
  Serum concentration of HDL cholesterol
LDL cholesterol | Baseline
  Serum Calculated LDL Cholesterol levels
LDL cholesterol | 12 weeks
  Serum Calculated LDL Cholesterol levels
Triglycerides | Baseline
  Serum Triglycerides levels
Triglycerides | 12 weeks
  Serum Triglycerides levels

SECONDARY OUTCOMES:
Weight | Baseline
  Weight status
Weight | 12 weeks
  Weight status
Fat mass | Baseline
  Fat mass in kg, measured by Bioimpedance
Fat mass | 12 weeks
  Fat mass in kg, measured by Bioimpedance
Hemoglobin | Baseline
  Hemoglobin measured as mg/dL
Hemoglobin | 12 weeks
  Hemoglobin measured as mg/dL
Hematocrit | Baseline
  Hematocrit (%)
Hematocrit | 12 weeks
  Hematocrit (%)
Physical Activity | Baseline
  Measured through the IPAQ questionnaire
Physical Activity | 12 weeks
  Measured through the IPAQ questionnaire
Blood pressure | Baseline
  Measured in the dominant arm (mmHg)
Blood pressure | 12 weeks
  Measured in the dominant arm (mmHg)
Dietary intake | Baseline
  FFQ from the SUN Study
Dietary intake | 12 weeks
  FFQ from the SUN Study

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Investigacion en Nutricion. Universidad de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No